CLINICAL TRIAL: NCT00446901
Title: Selenium and Prostate Cancer: Clinical Trial on Availability to Prostate Tissue and Effects on Gene Expression
Acronym: SePros
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: World Cancer Research Fund International (Other)
Responsible Party: Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WCRF 2004/21; CMO nr. 2007/003; SePros 2006/02; NL14694.091.07
Record Dates: First submitted 2007-03-12; First posted 2007-03-13 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2011-03

CONDITIONS: Prostatic Neoplasms; Prostate Cancer
Keywords: Prostate Cancer; Selenium; Chemoprevention; Gene expression
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Selenium
- Selenium (selenized yeast) (Experimental): Selenium (selenized yeast) tablets, 300 ug/day
  Interventions: Dietary Supplement: Selenium

INTERVENTIONS:
Dietary Supplement: Selenium — Selenized yeast, 300 ug/day
  Other Names: SelenoPrecise, PharmaNord

SUMMARY:
The aim of this study is to determine whether selenium supplementation leads to changes in selenium levels and gene expression profiles in prostate tissue.

DETAILED DESCRIPTION:
Rationale: Prostate cancer is a frequently observed malignancy in men, especially in elderly men. Besides diagnosis and treatment, also prevention of prostate cancer is an important point of interest to reduce the incidence and mortality of prostate cancer. Selenium is considered to be a promising chemopreventive agent for prostate cancer. Exact mechanisms of chemoprevention by selenium are not fully understood. However, it is expected that selenium (among other effects) directly affects gene expression in the prostate.

Objective: The aim of this study is to get insight into bioavailability of selenium in prostate tissue and changes of gene expression profiles that might be responsible for selenium-induced chemoprevention. To meet this objective, the relationship between dietary selenium intake and changes in gene expression profiles, tissue selenium levels and blood flow in prostate tissue will be examined.

Study design: The present study is designed as a double-blind, randomized and placebo-controlled intervention trial. Blood samples, toenails, questionnaires, MR images and surgical specimens will be collected to examine effects of selenium supplementation.

Study population: The study population will consist of 60 men, diagnosed with prostate cancer and scheduled for radical prostatectomy. Written informed consent will be obtained from each participant.

Intervention: Participants will receive 300 ug selenium / day or a placebo during 5 weeks prior to radical prostatectomy. Selenium will be supplemented in the form of selenized yeast tablets (SelenoPrecise, Pharma Nord).

Main study parameters: Levels of selenium in prostate tissue and changes in prostate gene expression profiles of participants supplemented with selenium or placebo, compared before and after the short intervention period, will be considered as the main parameters of the present study. Besides gene expression profiles in prostate tissue, also gene expression profiles of peripheral mononuclear cells (PBMC), levels of selenium in blood and toenails and blood flow and permeability of blood vessels of prostate tissue will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* male
* biopsy proven prostate cancer
* scheduled for radical prostatectomy

Exclusion Criteria:

* liver diseases (e.g. hepatitis)
* kidney diseases
* inflammatory bowel diseases
* use of dietary supplements containing selenium
* adjuvant therapy for prostate cancer (e.g. hormonal therapy, HIFU)
* previously or concurrent diagnosed with cancer, other than prostate cancer

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
selenium levels in prostate tissue | after 5 weeks of intervention with selenium or placebo
changes in gene expression profiles in prostate tissue | after 5 weeks of intervention with selenium or placebo

SECONDARY OUTCOMES:
changes in blood flow, vessel permeability and exocrine functionality | after 5 weeks of intervention with selenium or placebo
changes in gene expression profiles in blood cells | after 5 weeks of intervention with selenium or placebo

CONTACTS AND LOCATIONS:
Overall Officials: J.A. Witjes, Md PhD Prof, Study Chair — University Medical Center St Radboud; L.A.L.M. Kiemeney, PhD Prof, Study Chair — University Medical Center St Radboud; P. van 't Veer, PhD Prof, Study Chair — Wageningen University; L.A. Afman, PhD, Study Chair — Wageningen University
Locations (2):
- Netherlands (2):
  - University Medical Centre St Radboud, Nijmegen, Gelderland
  - Wageningen University, Wageningen, Gelderland